CLINICAL TRIAL: NCT06196463
Title: Erector Spinae Plane (ESP) Block for Pain Management in Juvenile Idiopathic Scoliosis Surgery: a Single-center, Randomized Controlled Trial
Brief Title: Erector Spinae Plane (ESP) Block in Juvenile Idiopathic Scoliosis Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 454/2023/Sper/IOR
Record Dates: First submitted 2023-12-12; First posted 2024-01-09 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Juvenile Idiopathic Scoliosis, Multiple Sites in Spine
Keywords: idiopathic scoliosis; spine surgery; ESP block; pain control
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: The Study is a prospective randomized controlled double blind trial, The enrolment will be made in accordance to a Random Number Generator Program. After signing the informed consent, verifying the inclusion and exclusion criteria and enrolling the patient, a progressive number will be assigned to each patient in the study.
Who Masked: Participant, Care Provider
Masking Description: The operating room anesthetist will only be informed that the patient to take care of, has been enrolled in the study, while a closed non-transparent envelope, containing the indication for the treatment or standard care, numbered progressively and corresponding to the randomization number of the patient, will be given to the anesthetist on call who will perform the anesthetic block or sham block. The operating room anesthetist who will manage the patient during the operation will not be made aware of the group to which the patient belongs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (AG+ESP) Group (Active Comparator): In AG+ ESP Group , the ESP block and the General anesthesia will be performed together in the same patient
  Interventions: Procedure: Erector spinale block (ESP block)
- AG Group (Sham Comparator): In AG Group the ESP block wont' be performed, but only a shamed block, realized through 4 skin puncture
  Interventions: Procedure: AG + sham block

INTERVENTIONS:
Procedure: Erector spinale block (ESP block) — The Study has the Objective to analyze the efficacy of the ESP block in spine Surgery (juvenile idiopathic scoliosis) to control perioperative pain
  Arms: (AG+ESP) Group
Procedure: AG + sham block — General anesthesia
  Arms: AG Group

SUMMARY:
The goal of this prospective controlled randomized clinical trial is to compare two intraoperative anesthetic patient management in Spinal surgery for idiopathic scoliosis. In particular in one Group of adolescent patients, the Erector Spinae (ESP) Block (an ultrasound-guided regional anesthesia technique) will be performed in addition to general anesthesia before surgical incision, while in the other Group the usual care (only General anesthesia, no Application of regional Block) will be applied. The fact that the ESP block acts on the dorsal branches of the spinal nerves, which innervate the paraspinal and vertebral muscles, makes this technique useful in the pain management of spine surgery. The main questions the study aims to answer are:

1. Verify if the pain measured in the two comparison groups in the first 24 postoperative hours is lower in the ESP Group.
2. Verify if the quantity of e.v opioid used intraoperatively, is lower in ESP Group
3. Verify if in ESP Group the Quantity of additional analgesics calculated by self-administered PCA doses of morphine (patient-controlled analgesia) in the first 24 hours postoperatively is lower than those administered in the usual care Group.
4. Verify if there are some differences between the two studied groups as regard the: Time to resume walking (expressed in hours from post-operative awakening); bowel movement recovery time (expressed in hours from post-operative awakening); Hospitalization time (expressed in days from the date of surgery until discharge).

DETAILED DESCRIPTION:
Spinal surgery for idiopathic scoliosis represents one of the most important post-operative pains in terms of severity and frequency. Perioperative locoregional analgesia can contribute to more effective control of perioperative pain. The Erector Spinae (ESP) Block is an interfascial block performed by identifying the erector spinae muscle (erector spinae muscle) lateral to the spine under ultrasound guidance. A needle is then advanced through the muscle until it makes contact with the transverse vertebral process. At this Point the anesthetic is injected generating a sensitive Block. The ESP block is a simpler procedure to perform than an epidural anesthesia with the advantage of reducing the risks of direct spinal damage, epidural hematoma and central nervous system infection. Before entering the operating theater and proceeding with induction and general anesthesia, patients will be placed in a prone, lateral or sitting position and a light sedation together with a local anesthesia of the skin will be performed to make the execution of the ESP block painless. The operator who will perform the anesthetic block or sham block will be different from the one who administer the anesthesia during surgery and awakes the patients. Therefore he/she will be blind to the kind of group which the patients belong to. The ESP block will be performed in patients in the intervention group ("AG+ESP") with 15 ml (2.5 mg/ml) of levobupivacaine bilaterally at the level of the IV-VI and X-XII thoracic vertebra (total dose 150mg). Patients in the placebo group ("AG group") will be given 4 subcutaneous injections with an ultrasound-guided technique of saline solution of 1 ml each bilaterally at the level of the IV-VI and X-XII thoracic vertebra. After having performed the block, all patients will be returned to the supine position and induction of general anesthesia and intubation will be carried out. The anesthetist who will manage the anesthesia during surgery will be unaware of the patient's group and will administer intraoperative opioids in relation to arterial pressure values and heart rate, while postoperative NSAID and opioids (administered through a patient controlled) will be given to the patients of both group in accordance to a designed and similar protocol. In the perioperative periods the total amount of analgesics and opioids, the level of patient pain measured with a VAS (Visual analogue score) score and other parameters like food intake, walking, time to first bowel movements and food intake will be recorded.

This prospective randomized controlled study performed on patient candidates to spinal surgery for juvenile idiopathic scoliosis, aims to verify the safety, efficacy and feasibility of the ESP block as a single injection compared to standard general anesthesia. Similar studies have analyzed the efficacy of ESP block in degenerative spine surgery, but this kind of block have not been studied in a randomized controlled trial since yet in juvenile idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* Elective indication for spine surgery for idiopathic scoliosis at the Spinal Surgery Department and Clinic 1 of the Rizzoli Orthopedic Institute.
* ASA Status 1 - 3
* BMI<32
* Expression of assent to informed consent

Exclusion Criteria:

* Patients who have previously undergone spinal procedures or surgery;
* Age under 14 years
* Patients on chronic opioid therapy (defined as the use of opioids continuously in the previous 3 months);
* Neuro-muscular pathologies;
* Allergy to drugs that are part of the study protocol;
* Cognitive deficit.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Average pain in the two comparison groups the end of surgery). | First 24 postoperative hours and in particular at 4-8-12-24 hour after surgery
  This average is analyzed via Visual Analogue Scale (VAS) in the first 24 postoperative hours. the VAS scale measures the extent of pain. The patient is asked to assign a score between 0 and 10 to the pain she is experiencing, considering 0 as no pain and 10 as maximum pain perceived.

SECONDARY OUTCOMES:
Quantity of opioid analgesics used intraoperatively | during surgery
  This quantity is calculated as average pro/kg of fentanyl and total dose and total dosage of remifentanil and maximum infusion rate at the same concentration
PCA (patient controlled analgesia) boluses of morphine administered and attempted by patients | the first 48 postoperative hours
  Patient controlled analgesia electronic pump permits to record all the attempted boluses
total dosage of morphine (total mg) received by the patient | the first 48 postoperative hours
  Patient controlled analgesia electronic pump permits to record the all dosage of administered morphine

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy